CLINICAL TRIAL: NCT03354065
Title: Inmediate Feeding Tolerance in Patients With Mild and Acute Biliary Pancreatitis vs Early Feeding
Brief Title: Inmediate Feeding Tolerance in Acute Pancreatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, David Esmer, head of the surgery service of Central Hospital, SLP, Mex, Hospital Central "Dr. Ignacio Morones Prieto"
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-15
Record Dates: First submitted 2017-10-27; First posted 2017-11-27 (Actual); Last update posted 2017-11-27 (Actual); Status verified 2017-11

CONDITIONS: Acute Pancreatitis Due to Gallstones
Keywords: pancreatitis; mild; biliary; referring
MeSH Terms: conditions — Pancreatitis; Lymphoma, Follicular

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: blinding of the evaluator to the study group blinding of patient to study hypothesis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early oral feeding (Active Comparator): TIME OF FEEDING. 48 hours after pancreatitis general management is started ( liquid diet)
  Interventions: Dietary Supplement: TIME OF FEEDING
- Immediate oral feeding (Experimental): TIME OF FEEDING: 8 hours of after pancreatitis general management is started (enteral formula)
  Interventions: Dietary Supplement: TIME OF FEEDING

INTERVENTIONS:
Dietary Supplement: TIME OF FEEDING — Liquid ( Re Feeding 8 h ) OR Enteral Feeding ( re feeding 48 h)

SUMMARY:
Objective: Determine tolerance of immediate oral intake (8 hours posterior to the beginning of treatment) against traditional management (early feeding at 48hr) in patients with mild acute pancreatitis of biliary origin.

Double blind, randomized clinical trial

DETAILED DESCRIPTION:
The investigators included patients 15 - 85 years old, any sex. Diagnosis of mild acute pancreatitis according to the Ranson, APACHE II and BISAP.

Signed infromed consent to participate in the study. All participants had a hepatic and biliary ultrasound to determine the biliary etiology.

The investigators excluded patients with pancreatitis of nonbiliary etiology, pregnant, severe pancreatitis, cholangitis or choledocholithiasis demonstrated during the hospital stay or with other comorbidities.

ELIGIBILITY:
Inclusion Criteria:

Patients older than 15 years.

* Patients with a diagnosis of mild acute pancreatitis biliary.
* Patients who agree to enter the protocol.

Exclusion Criteria:

* Patients managed at another institution.

  * Patients with a diagnosis of pancreatitis of non-biliary etiology.
  * Patients with heart disease or lung disease.
  * Patients with organic failure.
  * Patients with pregnancy.
  * Patients with cholangitis.

Ages: 15 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Pancreatitis reactivation after oral Feeding | Measures at 24hours after the begining of the oral intake
  Resurgence of characteristically epigastric tansfictive pain, irradiated to the left, upper quadrant region after beginning the oral intake, systemic inflammatory response syndrome ( C reactive protein) or Significant leucocyte elevation
Pancreatitis reactivation after oral Feeding | Measures at 48hours after the begining of the oral intake
  Resurgence of characteristically epigastric tansfictive pain, irradiated to the left, upper quadrant region after beginning the oral intake, systemic inflammatory response syndrome ( C reactive protein) or Significant leucocyte elevation

CONTACTS AND LOCATIONS:
Overall Officials: Juan F Hernandez, Study Chair — Postgraduate office at UASLP

IPD SHARING:
Plan to Share IPD: No